CLINICAL TRIAL: NCT05458453
Title: An Exploratory Study of Esketamine in Patients After Thoracoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Esketamine and thoracoscopic
Record Dates: First submitted 2022-07-01; First posted 2022-07-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2022-08

CONDITIONS: Esketamine; Thoracoscopic Surgery
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine arm (Experimental): Self-controlled intravenous analgesia pump was used for continuous injection, and it was prepared according to sufentanil 1.5ug/ml+ esketamine 0.75ug/ml+16mg ondansetron. After the operation, the analgesic pump was connected, and sufentanil 0.1ug/kg/h+ e sketamine 0.05mg/kg/h was pumped continuously for 24 hours. The continuous infusion of analgesia pump is (kg body weight/15) ml/h. (e.g. 60kg, pump speed 4ml/h, total amount 96ml).
  Interventions: Drug: Esketamine
- Sufentanil arm (No Intervention): Continuous pumping with self-controlled intravenous analgesia pump. According to sufentanil 1.5ug/ml+16mg ondansetron. At the end of the operation, connect the analgesic pump, and pump it with sufentanil at 0.1ug/kg/h for 24 hours. The continuous infusion of analgesia pump is (kg body weight/15) ml/h. (e.g. 60kg, pump speed 4ml/h, total amount 96ml).

INTERVENTIONS:
Drug: Esketamine — Self-controlled intravenous analgesia pump was used for continuous injection, and it was prepared according to sufentanil 1.5ug/ml+ esketamine 0.75ug/ml+16mg ondansetron. After the operation, the analgesic pump was connected, and sufentanil 0.1ug/kg/h+ esketamine 0.05mg/kg/h was pumped continuously for 24 hours. The continuous infusion of analgesia pump is (kg body weight/15) ml/h. (e.g. 60kg, pump speed 4ml/h, total amount 96ml).
  Arms: Esketamine arm

SUMMARY:
Thoracic surgery can produce severe postoperative acute pain, which can easily lead to cough weakness, atelectasis, respiratory restriction, pneumonia, hypoxemia, secretion retention, respiratory failure and other adverse events. Esketamine can reduce the demand of analgesic opioids, reduce the respiratory depression caused by opioids, improve ventilation, significantly reduce postoperative pain and prolong the analgesic time after thoracic surgery. Therefore, the application of esketamine in postoperative analgesia of patients undergoing thoracoscopic surgery may help to improve the respiratory function of clinical patients and further improve the postoperative analgesia effect, so as to achieve the purpose of accelerating the surgical rehabilitation of patients undergoing thoracoscopic surgery. Esketamine is rarely used in perioperative period in China, and the development of its safe and reasonable application methods and potential role in perioperative anesthesia needs further research and verification. Generally speaking, at present, there is still a lack of evaluation of ketamine in improving respiratory function, pain, anxiety and depression after thoracoscopic surgery, and there is no direct clinical evidence.

At present, sufentanil is the most commonly used drug for postoperative analgesia in patients undergoing clinical surgery. As a strong opioid, although sufentanil can provide good analgesic effect, the respiratory depression caused by sufentanil is not conducive to the recovery of postoperative lung function in patients undergoing thoracic surgery. The action sites of esketamine include N- methyl-aspartic acid (NMDA) receptor, opioid receptor, monoamine receptor, M cholinergic receptor, sodium channel, calcium channel, etc., which can relieve respiratory depression caused by opioids, stimulate respiration, relax airway smooth muscle, prevent hyperalgesia caused by opioids, reduce the dosage of postoperative analgesics and prolong the duration of postoperative analgesia. Therefore, esketamine is likely to improve postoperative respiratory function of patients after thoracoscopic surgery and play a good role. To sum up, this study is intended to include patients undergoing elective thoracoscopic surgery. Through a prospective randomized controlled double-blind clinical trial, different analgesic drugs of intravenous patient-controlled analgesia and simple conventional opioid analgesic sufentanil are used as the control. Combined with the investigation of preoperative and postoperative tidal volume, oxygenation index, postoperative pain and postoperative recovery outcome, the effects of esketamine on postoperative respiratory function, postoperative pain and overall rehabilitation of these patients are compared, so as to provide direct clinical evidence for improving postoperative lung function of patients undergoing elective thoracoscopic surgery, and at the same time, provide a choice for thoracoscopic surgery.

To explore the effect of esketamine on improving postoperative respiratory function, pain, depression and anxiety and overall rehabilitation of patients undergoing thoracoscopic surgery. Compound esketamine is used for postoperative analgesia, thus providing direct clinical evidence for improving postoperative pulmonary function of patients undergoing elective thoracoscopic surgery, and providing reference for improving postoperative pain, anxiety and depression of patients undergoing elective thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing thoracoscopic surgery are required to use PCIA for analgesia;
2. ASA grade I-III;
3. The patient's age is 18-75 years old; 4、18.5 < BMI < 28；

5. Obtain the informed consent of patients and their families;

Exclusion Criteria:

1. Patients with previous history of thoracic surgery or combined history of thoracic trauma;
2. Patients with severe hypertension and poor control;
3. Patients with hyperthyroidism and poor control;
4. Patients at risk of increased intracranial pressure;
5. Patients with mental illness;
6. Patients who are allergic to any drug in the test;
7. Patients who take anti-inflammatory drugs, opioids or related diseases for a long time;
8. Pregnant or lactating patients;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Minute ventilation volume 0 | Before anesthesia induction
  Minute ventilation volume before anesthesia induction
Minute ventilation volume 1 | Within 5 minutes after extubation
  Minute ventilation volume after extubation
Minute ventilation volume 2 | postoperative day 1 (POD1) morning
  Minute ventilation volume on the first morning
Minute ventilation volume 3 | postoperative day 1 (POD1) afternoon
  Minute ventilation volume on the first afternoon
Minute ventilation volume 4 | postoperative day 2 (POD2) morning
  Minute ventilation volume on the next morning
Minute ventilation volume 5 | postoperative day 2 (POD2) afternoon
  Minute ventilation volume on the next afternoon
Tidal volume 0 | Before anesthesia induction
  Tidal volume before anesthesia induction
Tidal volume 1 | Within 5 minutes after extubation
  Tidal volume after extubation
Tidal volume 2 | Day1 （The first morning after surgery）
  Tidal volume on the first morning after surgery
Tidal volume 3 | Day1（The afternoon of the first day after surgery）
  Tidal volume on the first afternoon after surgery
Tidal volume 4 | day 2 ( second morning after surgery)
  Tidal volume on the next morning after surgery
Tidal volume 5 | day 2 ( second afternoon after surgery)
  Tidal volume on the next afternoon after surgery
Respiratory rate 0 | Before anesthesia induction
  Respiratory rate before anesthesia induction
Respiratory rate 1 | Within 5 minutes after extubation
  Respiratory rate after extubation
Respiratory rate 2 | Day1 （The first morning after surgery）
  Respiratory rate on the first morning after surgery
Respiratory rate 3 | Day1 （The afternoon of the first day after surgery）
  Respiratory rate on the first afternoon after surgery
Respiratory rate 4 | day 2 ( second morning after using surgery)
  Respiratory rate on the next morning after surgery
Respiratory rate 5 | day 2 ( second afternoon after surgery)
  Respiratory rate on the next afternoon after surgery

SECONDARY OUTCOMES:
Vas score 1 | Within 5 minutes after extubation
  The higher the score, the more painful it is.
Vas score 2 | postoperative day 1 (POD1) morning
  The higher the score, the more painful it is.
Vas score 3 | postoperative day 1 (POD1) afternoon
  The higher the score, the more painful it is.
Vas score 4 | postoperative day 2 (POD2) morning
  The higher the score, the more painful it is.
Vas score 5 | postoperative day 2 (POD2) afternoon
  The higher the score, the more painful it is.
Oxygenation index 0 | Before anesthesia induction
  Oxygenation index (calculated as PaO2/FiO2) before anesthesia induction
Oxygenation index 1 | Within 5 minutes after extubation
  Oxygenation index (calculated as PaO2/FiO2) after extubation
Oxygenation index 3 | postoperative Day 1
  Oxygenation index (calculated as PaO2/FiO2) on the first morning
Incidence of postoperative pulmonary complications during hospitalization | From end of the surgery to hospital discharge with about mean of 7 days after surgery
  postoperative pulmonary complications during hospitalization was assessed using the Melbourne Group Scale, whcih reached four or more of the 8 criteria would be diagnosed with postoperative pulmonary complications.
incidence of hypoxemia during the first and second day after surgery | from end of the surgery to the second day after surgery
  hypoxemia is defined as SpO2<92% during the first and second day after surgery

OTHER OUTCOMES:
Depression scale 0 | Before anesthesia induction
  PHQ-9， The higher the score, the more depressed.
Depression scale 2 | Day 1(the first morning after using PCIA)
  PHQ-9，The higher the score, the more depressed.
Depression scale 4 | day 2 ( second morning after using PCIA)
  PHQ-9，The higher the score, the more depressed.
anxiety score 0 | Before anesthesia induction
  GAD-7，The higher the score, the more anxious.
anxiety score 2 | Day1(the first morning after using PCIA)
  GAD-7，The higher the score, the more anxious.
anxiety score 4 | day 2 ( second morning after using PCIA)
  GAD-7，The higher the score, the more anxious.
sleep quality during the first two days after surgery | from end of the surgery to the second day after surgery
  assessed by Richards-Campbell sleep score, which higher socre represents better sleep quality

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year

REFERENCES:
- [Derived] Fu M, Xu R, Chen G, Zheng X, Shu B, Huang H, Duan G, Chen Y. Postoperative esketamine improves ventilation after video-assisted thoracoscopic lung resection: A double-blinded randomized controlled trial. Heliyon. 2024 Jan 24;10(3):e25100. doi: 10.1016/j.heliyon.2024.e25100. eCollection 2024 Feb 15. PMID 38322862